CLINICAL TRIAL: NCT05754970
Title: Clinical, Prospective, Non-profit, Non-pharmacological Study on Geass Healing Abutment: Microbiological, Histological, and Immuno-histochemical Evaluation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Professor, G. d'Annunzio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2218102018
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Intervention Model Description: To prevent allocation bias among patients, each healing abutment was designed with two surfaces that alternated between laser-treated/machined and ma-chined/laser-treated. The experimental healing abutment was removed after 30 ± 7 days, which coincided with the soft tissue biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laser/machined (Experimental): on the same customized healing abutment laser-treated/machined surface treatments were repeated with the following order: Laser treated/machined/laser treated/machined. This order was performed to eliminate the bias of the different surface allocation on patients.
  Interventions: Procedure: laser treated

INTERVENTIONS:
Procedure: laser treated — The second surgical stage was done after a healing period 12 ± 4 weeks (T1) where all the healing abutments were placed. Each healing abutment had repeated the two surfaces as twice follows: laser-treated/machined/ laser-treated/machined. Experimental healing abutment was removed after 30 ± 7 days, the same time as the soft tissue biopsy.
  After the healing period (30 ± 7 days), before starting with the prosthetic restoration of the fixtures, an impression was taken of the small-diameter Has, and circular sections (diameter 5 mm) soft tissues around them were retrieved for analysis.

SUMMARY:
The health of peri-implant soft tissues is important for the long-term success rate of dental implants and the surface topography is pivotal in influencing it. Thus, the aim of this study was to evaluate, in human patients, the inflammatory mucosal microenvironment in the tissue surrounding a new, nanoscale, laser-treated healing abutment characterized by engineered nanopores versus a standard machined-surface.

The prospective clinical study will evaluate the effect of the presence of a laser-etched surface in the coronal portion of healing stumps in forming the coronal seal and reducing the accumulation of bacterial plaque around it. The screws will serve as their own control group since they have both a laser-etched and a smooth portion.

Primary objective:

To evaluate the adhesion of fibroblastic cells from the peri-implant mucosa on the surface of the healing stump through scanning electron microscope analysis, expressed in terms of the area covered by the cells.

Secondary objectives:

To evaluate the amount of bacterial adhesion around healing stumps with a laser-etched and smooth altered surface through scanning electron microscope analysis, expressed in terms of the area covered by the cells.

To evaluate the presence of hemidesmosomal structures through the expression of α-6 and β-4 integrins.

To evaluate bacterial adhesion on healing screws. To evaluate the healing of peri-implant soft tissues through clinical indices, such as Plaque Index and Gingival Index.

The healing period was 12 ± 4 weeks (T1) before the second surgical procedure, during which all healing abutments were placed. To prevent allocation bias among patients, each healing abutment was designed with two surfaces that alternated between laser-treated/machined and ma-chined/laser-treated. The experimental healing abutment was removed after 30 ± 7 days, which coincided with the soft tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years
* Patients with no systemic and/or oral health disease
* At least six months of healing after tooth extraction
* Adequate dimension of the attached gingiva (>2 mm) or keratinized tissue at the site selected and adequate residual bone crest

Exclusion Criteria:

* - Patients with poor oral hygiene
* Plaque score (PS) and bleeding on probing (BOP) more than 25%
* Patients with active periodontal disease
* Insufficient bone thickness for implant insertion and bone augmentation procedures
* patients who necessitate immediate implant loading protocols
* Uncontrolled diabetes mellitus
* Immune diseases
* Patients who smoke more than 10 cig/die

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
soft tissue adhesion | After a healing period of 12 ± 4 weeks, during the second surgical phase
  To evaluate the adhesion of fibroblastic cells from the peri-implant mucosa on the surface of the healing stump through scanning electron microscope analysis, expressed in terms of the area covered by the cells.

SECONDARY OUTCOMES:
bacterial adhesion | After a healing period of 12 ± 4 weeks, during the second surgical phase
  To evaluate the amount of bacterial adhesion around healing stumps with a laser-etched and smooth altered surface through scanning electron microscope analysis, expressed in terms of the area covered by the cells.

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belloni A, Argentieri G, Orilisi G, Notarstefano V, Giorgini E, D'Addazio G, Orsini G, Caputi S, Sinjari B. New insights on collagen structural organization and spatial distribution around dental implants: a comparison between machined and laser-treated surfaces. J Transl Med. 2024 Jan 31;22(1):120. doi: 10.1186/s12967-024-04906-4. PMID 38297308
- [Derived] Gaggi G, Di Credico A, D'Addazio G, Ghinassi B, Argentieri G, Caputi S, Di Baldassarre A, Sinjari B. Impact on peri-implant connective tissue of laser treated versus traditional healing abutments: a human clinical trials. BMC Oral Health. 2023 Jun 27;23(1):425. doi: 10.1186/s12903-023-03148-y. PMID 37370064